CLINICAL TRIAL: NCT06064799
Title: Expression of microRNA-223 and microRNA-214 in Gingival Crevicular Fluid of Smoker and Nonsmoker Periodontitis Patients, an Observational Diagnostic Accuracy Study
Brief Title: GCF miRNA-223 , -214 Levels in Smokers and Nonsmokers Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Nayroz Tarrad, associate professor, Fayoum University
Other Study IDs: REC-FDBSU/05012023-04/AM
Record Dates: First submitted 2023-09-20; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis, Adult
Keywords: Periodontitis; microRNA; smoking; GCF; biofluids
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — GCF samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: 14 healthy volunteers
  Interventions: Diagnostic Test: miRNA-223 & -214 detection
- Group II: 14 periodontitis participants with stage III grade B Periodontitis
  Interventions: Diagnostic Test: miRNA-223 & -214 detection
- Group III: 14 periodontitis participants with stage III grade C Periodontitis
  Interventions: Diagnostic Test: miRNA-223 & -214 detection

INTERVENTIONS:
Diagnostic Test: miRNA-223 & -214 detection — miRNA-223 & -214 detection in GCF samples by PCR kits

SUMMARY:
Objective: Periodontitis is a multifactorial disease that affects a wide range of populations. However, its pathogenesis remains unclear. miRNAs are now considered potential diagnostic markers for many inflammatory diseases. Thus, the aim of this study was to assess the expression of microRNA-223(miRNA-223) and microRNA-214 (miRNA-214) in gingival crevicular fluid (GCF) of smoker and nonsmoker with periodontitis.

Materials and Methods: We conducted a prospective study among 42 participants: 14 healthy controls, 14 nonsmoker periodontitis participants, and 14 smoker with periodontitis. Eligibility criteria for inclusion were consecutive adults, aged 20-60 years, with stage III periodontitis grade B/C and no systemic diseases. All consenting participants had gingival crevicular fluid samples collected after diagnosis to assess miRNA-214 and -223 by quantitative real-time polymerase chain reaction assay.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* age from 20 to 60 years
* no more than 4 teeth lost due to periodontitis
* systemically free participants

Exclusion Criteria:

* Pregnant or lactating female
* participants with a history of an inflammatory or immunological disease
* history of any current medication

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: individuals were recruited from the outpatient clinic of the department of periodontology
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
assessment of miRNA-223 & -214 levels in GCF samples in all groups | level of miR-223 & -214 are measured at baseline after the completion of all GCF sample collection carried at the day of enrollment of subjects in the investigation after diagnosis confirmation
  PCR kits are used for assessment of miRNA-223 & -214 levels in GCF samples in all groups

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Fayoum university, Al Fayyum, Egypt